CLINICAL TRIAL: NCT06991140
Title: Investigation of the Efficacy of Thoracic Mobilization Exercises Performed in Addition to Core Stabilization Exercises in Individuals With Chronic Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758)
Record Dates: First submitted 2025-05-15; First posted 2025-05-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain
Keywords: neck pain; mobilization
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Core stabilisation exercises applied to both groups of the study were structured to target the activation of deep muscle groups supporting the stability of the cervical and thoracic spine. The exercise programme was performed 3 days a week for a total of 6 weeks under the supervision of a physiotherapist. The programme included exercises to improve head and neck control (chin tuck, head lift in supine position), exercises to improve scapular stability (scapular retraction, wall slide, serratus anterior activation) and exercises to improve trunk control in neutral spine position (arm and leg extension in four-point position, plank variations). The exercises were gradually made more difficult according to the tolerance of the individuals and each session lasted approximately 40-45 minutes. By ensuring that the exercises were performed in the correct form and in a controlled manner, overloading of the musculoskeletal system was prevented.
  Interventions: Other: Core Stabilization Exercises
- Thorocal mobilization group (Experimental): Thoracic mobilisation exercises were performed 3 days a week for a total of 6 weeks under the supervision of a physiotherapist. Thoracic mobilisation programme consisted of active self-mobilisation techniques, mobilisation exercises with foam rollers, stretching exercises including thoracic rotation and extension movements and dynamic postural exercises. Especially 'thread the needle' exercise in sitting or quadruped position, 'thoracic extension press-up' in prone position and 'extension on foam rollers' were preferred to increase the mobility of thoracic vertebral segments. The exercises were gradually made more difficult according to the tolerance of the individuals. Each exercise was performed as 10-15 repetitions and 2-3 sets. Exercise safety was ensured by informing the patients about the correct posture and movement patterns before all applications. The main aim of the exercises was to alleviate the mechanical load of the cervicothoracic transition by reducing thoracic hypomobi
  Interventions: Other: Thorocal Mobilization Exercises; Other: Core Stabilization Exercises

INTERVENTIONS:
Other: Thorocal Mobilization Exercises — Thoracic mobilisation exercises were performed 3 days a week for a total of 6 weeks under the supervision of a physiotherapist. Thoracic mobilisation programme consisted of active self-mobilisation techniques, mobilisation exercises with foam rollers, stretching exercises including thoracic rotation and extension movements and dynamic postural exercises. Especially 'thread the needle' exercise in sitting or quadruped position, 'thoracic extension press-up' in prone position and 'extension on foam rollers' were preferred to increase the mobility of thoracic vertebral segments. The exercises were gradually made more difficult according to the tolerance of the individuals. Each exercise was performed as 10-15 repetitions and 2-3 sets. Exercise safety was ensured by informing the patients about the correct posture and movement patterns before all applications.
  Arms: Thorocal mobilization group
Other: Core Stabilization Exercises — Core stabilization exercises were structured to target activation of deep muscle groups supporting cervical and thoracic spine stability. The exercise programme was performed 3 days a week for a total of 6 weeks under the supervision of a physiotherapist. The programme included exercises to improve head and neck control (chin tuck, head lift in supine position), exercises to improve scapular stability (scapular retraction, wall slide, serratus anterior activation) and exercises to improve trunk control in neutral spine position (arm and leg extension in four-point position, plank variations). The exercises were gradually made more difficult according to the tolerance of the individuals and each session lasted approximately 40-45 minutes. By ensuring that the exercises were performed in the correct form and in a controlled manner, overloading of the musculoskeletal system was prevented.

SUMMARY:
Neck pain is one of the most common musculoskeletal complaints worldwide and is an important health problem that restricts the daily life activities of individuals. In particular, chronic non-specific neck pain (CNSNP) describes pain that persists for at least 12 weeks without an underlying specific pathological cause and affects a large segment of the population. CNSNP leads not only to pain but also to functional limitations, postural disorders and decreased quality of life.

In recent years, exercise-based approaches, especially core stabilisation exercises, have become prominent in the treatment of CNSNP. Core stabilisation exercises aim to increase postural control, improve segmental stability and thus reduce pain by activating deep muscle groups around the spine. However, it has been reported that exercises targeting only local muscle groups may be insufficient to meet the high-level biomechanical and neuromuscular needs of the cervical spine.

In this context, the effect of the mobility of the thoracic spine on neck function is noteworthy. Hypomobility in the thoracic region may contribute to pain and dysfunction by increasing the load on the cervical spine. Therefore, it is thought that adding thoracic mobilisation exercises to core stabilisation exercises may be more effective in improving neck pain and postural disorders.

The aim of this study was to investigate the effects of adding thoracic mobilisation to a core stabilisation exercise programme in individuals with chronic non-specific neck pain.

DETAILED DESCRIPTION:
Neck pain is one of the most common musculoskeletal problems on a global scale and causes a significant decrease in the quality of life by negatively affecting the social, occupational and physical functionality of individuals. It is reported that approximately 30-50% of individuals experience neck pain every year and a significant proportion of these complaints become chronic. Chronic non-specific neck pain (CNSNP) is defined as neck pain that persists for more than three months without an underlying anatomical or pathological cause and is the most common type of neck pain encountered in clinical practice. In the treatment of CNSNP, both symptom relief and correction of underlying mechanical disorders are important.

In rehabilitation programmes for neck pain, core stabilisation exercises are widely used to strengthen spinal stability and improve postural control by increasing activation of the deep muscles supporting the cervical and thoracic spine. The core consists of a large number of muscles and connective tissues surrounding the lumbar, thoracic and cervical spine and the coordinated functioning of these structures is critical for the functional integrity of the spine. Various studies have shown that core stabilisation exercises are effective in reducing pain and increasing functional capacity.

However, the functional and mechanical health of the cervical spine is closely related not only to the local stabilising muscles but also to the mobility of the thoracic spine. Hypomobility of the thoracic spine can lead to increased compensatory motion in the cervical segments, muscle spasm, postural distortion and increased pain. There is increasing evidence in the literature that improving thoracic mobility can reduce cervical pain and dysfunction. In this context, integrating thoracic mobilisation exercises into core stabilisation programmes may provide not only symptomatic relief, but also better postural alignment and more effective functional recovery.

The aim of this study is to comparatively examine the effects of adding thoracic mobilisation exercises to core stabilisation exercises in individuals with chronic non-specific neck pain. In this direction, it is aimed to evaluate the extent to which the applications for the mobility of the thoracic spine affect the clinical symptoms in the cervical region and to obtain data that will contribute to clinical rehabilitation programmes.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65,
* 3 months of persistent neck pain,
* Being sedentary,
* Not being involved in any physiotherapy programme in the last 6 months

Exclusion Criteria:

* History of previous spinal surgery or trauma,
* Neurological deficit, vestibular pathology, neurological, cardiopulmonary, musculoskeletal problems affecting physical performance, any pathology in the shoulder joint, any pathology in the jaw joint and pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 6 week
  Visual Analogue Scale was used to determine severity of low back pain in the study participants. Visual Analogue Scale is a practical test with high validity and reliability in pain assessment. Visual Analogue Scale is an assessment method numbered from 0 to 10, where '0' indicates no pain and '10' indicates the presence of the most severe pain. Participants were asked to mark the degree of pain they had on this scale and recorded.

SECONDARY OUTCOMES:
Disability | 6 week
  The Neck Disability Index consists of 10 headings. Participants are asked to score each question between 0 (no disability) and 5 (full disability). The total score ranges from 0 (no disability) to 50 (total disability). A score of 0-4 is interpreted as no disability, 5-14 as mild disability, 15-24 as moderate disability, 25-34 as severe disability and >35 as total disability.
Cervical muscle strength | 6 week
  Flexor and extensor muscle strength of the cervical region was measured with a digital hand dynamometer (Lafayette Instrument Company, USA). For the evaluation position, the fine muscle test positions and method defined by Lovett were taken as a basis. While evaluating the cervical flexors, participants were asked to flex their heads while lying in the supine position in the hook position, and the resistance was given from the frontal region. While evaluating the cervical extensors, participants were asked to extend their heads in the prone position with the arms at their sides, the resistance was given from the occipital region. All measurements were repeated three times and the highest value was recorded in kilogram.
Spine Assessment | 6 week
  Spine structure was assessed with the Spinal Mouse® (Idiag, Volkerswill, Switzerland) device . It is a non-invasive, radiation-free, and computer-assisted electromechanical device. The handheld wireless mouse included in the device is connected to a computer via bluetooth. The raw data reaches the computer via bluetooth and is evaluated by the software. The device has measurement options in different planes, provides the opportunity to evaluate both the posture and mobility of the spine, and gives valid, and reliable results. During the assessment, the processes spinosus of the spine from C7 to S3 were marked and the mouse was slide along the spine from top to bottom from the skin surface at a constant speed and pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, PhD., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No